CLINICAL TRIAL: NCT03927768
Title: Abbreviated Breast MRI (AB-MRI) With Golden-angle Radial Compressed-sensing and Parallel Imaging (GRASP): a Short, Comprehensive Breast MRI Exam Ready for Clinical Prime Time.
Brief Title: Abbreviated Breast MRI (AB-MRI) With Golden-angle Radial Compressed-sensing and Parallel Imaging (GRASP)
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-00684
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Predictive Learning Models

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 200 women undergoing clinical breast MRI: At time of previously scheduled clinical breast MRI, 60 second postcontrast imaging sequence will be added to the clinical breast MRI. MRI will be interpreted according to usual departmental protocols.
  Interventions: Diagnostic Test: Predictive Model; Diagnostic Test: Breast Imagers
- 50 women undergoing clinical breast MRI: At time of previously scheduled clinical breast MRI, 60 second postcontrast imaging sequence will be added to the clinical breast MRI. MRI will be interpreted according to usual departmental protocols.
  Interventions: Diagnostic Test: Predictive Model; Diagnostic Test: Breast Imagers

INTERVENTIONS:
Diagnostic Test: Predictive Model — Anonymized, post-processed MRI imaging data will be analyzed to construct a model predicting benign vs malignant lesions. Model will be tested on a second cohort.
Diagnostic Test: Breast Imagers — Anonymized research sequence with the addition of modeling data (Aims 1A and 1B) will be read by three blinded breast imagers and final evaluation compared to the full protocol.

SUMMARY:
The purpose of this study is to use a magnetic resonance imaging (MRI) sequence called golden-angle radial compressed sensing and parallel imaging (GRASP) as a noninvasive and fast way to measure the wash-in contrast (dye) in the breast. MRI uses a strong magnetic field and radio waves to create images of structures in the body. The goal is to determine if benign and malignant breast lesions have different patterns of contrast wash in.

This study will ask woman planning to undergo a clinical breast MRI with contrast (dye) as part of their standard care.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications to MRI scanning (pacemaker, implanted metallic objects, severe obesity or other condition that leads to difficulty lying in the magnet)
* Able and willing to provide informed consent

Exclusion Criteria:

* Currently undergoing neoadjuvant chemotherapy for breast cancer treatment.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 women scheduled for clinical breast MRI
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic accuracy of GRASP AB-MRI temporal kinetics in the diagnosis of breast malignancies. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Heacock, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication
Access Criteria: Requests may be directed to the PI